CLINICAL TRIAL: NCT03930511
Title: Impact of Pulmonary Rehabilitation on Physical Activity in Daily Life on Chronic Respiratory Patients - SmartReab Telemonitoring
Brief Title: Telemonitoring Physical Activity in Daily Life on Chronic Respiratory Patients
Acronym: SmartReab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Collaborators: Centro Hospitalar Lisboa Norte (Other); CAST - Consultoria e Aplicações em Sistemas e Tecnologia, Lda. (Unknown); Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Catarina Santos, PhD student, Physiotherapist MSc, University of Lisbon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 02/17
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Chronic Respiratory Disease
Keywords: Telemonitoring; Physical activity; Pulmonary Rehabilitation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PADL at the beginning of PR (No Intervention): First assessment of patients starting Pulmonary Rehabilitation, including a 4 day time telemonitoring of physical activity on daily life, 6 minute walk test, International Physical Activity Questionnaire (IPAQ), EuroQoL, mMRC, COPD Assessment Test (CAT), London Chest Activity of Daily Living (LCADL) and Hospital Anxiety and Depression Scale (HADS).
- PADL at discharge of PR (Experimental): Assessment of patients at discharge of Pulmonary Rehabilitation, including a 4 day time telemonitoring of physical activity on daily life, 6 minute walk test, International Physical Activity Questionnaire (IPAQ), EuroQoL, mMRC, COPD Assessment Test (CAT), London Chest Activity of Daily Living (LCADL) and Hospital Anxiety and Depression Scale (HADS).
  Interventions: Procedure: Pulmonary Rehabilitation
- PADL at 6 months follow-up (No Intervention): Half-a-year reassessment of patients on Pulmonary Rehabilitation, including a 4 day time telemonitoring of physical activity on daily life, 6 minute walk test, International Physical Activity Questionnaire (IPAQ), EuroQoL, mMRC, COPD Assessment Test (CAT), London Chest Activity of Daily Living (LCADL) and Hospital Anxiety and Depression Scale (HADS).
- PADL at 1 year follow-up (No Intervention): Yearly reassessment of patients on Pulmonary Rehabilitation, including a 4 day time telemonitoring of physical activity on daily life, 6 minute walk test, International Physical Activity Questionnaire (IPAQ), EuroQoL, mMRC, COPD Assessment Test (CAT), London Chest Activity of Daily Living (LCADL) and Hospital Anxiety and Depression Scale (HADS).

INTERVENTIONS:
Procedure: Pulmonary Rehabilitation — According to patients' needs and physician referral, individually tailored treatments of respiratory physiotherapy, functional training, exercise training and patient education
  Arms: PADL at discharge of PR

SUMMARY:
Physical inactivity is a consequence of chronic diseases and on Chronic Obstructive Pulmonary Disease patients is an independent predictor of the risk of hospitalizations and early mortality. As physical inactivity is a modifiable risk factor with healthy lifestyle interventions, health professionals should clinically assess physical activity as a vital sign of patients' general physical condition. SmartReab study aims to characterize physical activity in daily life of 100 chronic respiratory patients at baseline when starting Pulmonary Rehabilitation, at discharge time of the program, at 6 months and 1 year follow-up. The Pulmonary Rehabilitation program will be individually tailored according to patients needs and goals settled within the Rehabilitation team and it will take place at Hospital Pulido Valente, from Centro Hospitalar Universitário Lisboa Norte, in Lisbon, Portugal. To access physical activity in daily life patients will participate in a telemonitoring study for 4 days using a smartphone and an oximeter and also answer to the International Physical Activity Questionnaire. SmartReab technology will provide data of physical activity intensity, heart rate and oxygen levels during awakening periods of daytime. To associate physical activity with other aspects related with health and the impact of Pulmonary Rehabilitation, patients will also take a 6 minute walk test and answer questionnaires related with self-perceived health status, impact of respiratory symptoms on quality of life, dyspnea impact on general mobility and on daily life situations, and also anxiety and depression feelings. The research hypothesis is that Pulmonary Rehabilitation will have a positive impact on physical activity in the short, medium and long terms.

DETAILED DESCRIPTION:
The Global Alliance Against Chronic Respiratory Diseases (GARD) stated physical inactivity as a modifiable risk factor for all chronic respiratory diseases and advocates stakeholders for action, including the health care community. With respect to chronic respiratory conditions, evidence on Chronic Obstructive Pulmonary Disease indicates physical inactivity as an independent predictor of the risk of hospitalizations due to acute exacerbations and untimely mortality. Exercise is Medicine® is an initiative of the American College of Sports Medicine which encourages all health care professionals to promptly assess physical activity habits as a vital sign of general physical condition, optimizing exercise counselling or referral and enhancing chronic disease management. Because of this, research directions on Pulmonary Rehabilitation target on methodology development for physical activity assessment, combining subjective patient reported experience and accurate objective measurement on patients' daily life. Hospital Pulido Valente in Lisbon, Portugal, started TELEMOLD, which developed an Android smartphone telemonitoring system with a mobile software application connected to an oximeter and accelerometer sensors. Presently the project evolved to SMARTREAB applying such technology to a combined assessment of pulse oximetry and physical activity as a routine procedure with respiratory patients. This study aims to characterize baseline physical activity in daily life of 100 chronic respiratory patients on Pulmonary Rehabilitation as a primary endpoint. Secondary endpoints include reassessments of physical activity in daily life at discharge from the program, 6 months and 1 year follow-up. The Pulmonary Rehabilitation program will be individually tailored according to patients needs and goals settled within the Rehabilitation team and it will take place at Hospital Pulido Valente, from Centro Hospitalar Universitário Lisboa Norte, in Lisbon, Portugal. Patients' assessments include a 4 days SmartReab telemonitoring study providing data of physical activity intensity, heart rate and oxygen levels during awakening periods of daytime. Patients will further participate in a 6 minute walk test and answer selected questionnaires: the International Physical Activity Questionnaire (IPAQ) , the visual analogue scale of the EuroQoL (EuroQoL-VAS), the modified Medical Research Council dyspnea scale (mMRC), the COPD assessment test (CAT), the London Chest Activity of Daily Living scale (LCADL) and the Hospital Anxiety and Depression Scale (HADS). The research hypothesis is that Pulmonary Rehabilitation will have a positive impact on physical activity in the short, medium and long terms in association with other secondary outcomes assessed. All patients gave informed consent and ethical approval was obtained by the Ethics Committee of Centro Hospitalar Universitário Lisboa Norte, EPE and Centro Académico de Medicina de Lisboa (number 02/17). Statistical analysis will be performed using the Statistical Package for the Social Sciences (SPSS) version 25.0 (SPSS Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* chronic lung disease
* patient referenced to Pulmonary Rehabilitation

Exclusion Criteria:

* pleural effusion
* infectious disease
* unstable cardiac disease
* neurologic or musculoskeletal conditions affecting exercise performance
* cognitive deficit affecting questionnaire comprehensive answer
* psychiatric disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Objective Physical Activity in Daily Life | 4 days excluding night sleeping
  Percentage of time spent (0-100%) on three categories of physical activity measured as metabolic equivalent of task (MET) by telemonitoring with an accelerometer incorporated in a smartphone: less than 2 MET, between 2 and 3 MET, above 3 MET.
Reported Physical Activity in Daily Life | 1 week
  METS per week as answered to the International Physical Activity Questionnaire considering the domains of work, transport, domestic and gardening, and leisure time; additional data for reported sedentary time with sitting time per week

SECONDARY OUTCOMES:
Functional capacity | 6 minutes
  distance (meters) on the 6 minute walk test
Perceived general health | 1 day
  EuroQoL visual analogue scale (0-100) of perceived general health
Perceived dyspnea | 1 day
  modified Medical Research Council scale graduating perceived dyspnea from 0 to 4, with higher values associated to increased dyspnea on minimal activities
Symptoms impact on quality of life | 1 day
  COPD Assessment Test (CAT) score (0-40) with higher values associated to greater impact of respiratory disease symptoms on quality of life
Perceived dyspnea on daily activities | 1 day
  London Chest Activity of Daily Living (LCADL) scale score (0-75) assessing on a scale from 0-5 (with higher values indicating increased limitation or dependency) subscores of self-care (0-20), domestic (0-30), social (0-15) and physical activities (0-10)
Anxiety and Depression | 1 week
  Hospital Anxiety and Depression Scale (HADS) assessing on a scale from 0-3, seven questions about anxiety and seven questions about depression; score is reported ranging from 0-21 separately to depression and anxiety; higher values are associated with increased anxiety/depression

CONTACTS AND LOCATIONS:
Overall Officials: Catarina D Santos, MSc, Principal Investigator — University of Lisbon; Cristina Bárbara, PhD, Study Director — University of Lisbon
Locations (2):
- Portugal (2):
  - Universidade de Lisboa, Faculdade de Medicina, Instituto de Saúde Ambiental (ISAMB), Lisbon
  - CAST - Consultoria e Aplicações em Sistemas e Tecnologia, Lda., Lisbon

IPD SHARING:
Plan to Share IPD: No